CLINICAL TRIAL: NCT00471653
Title: A Pharmacokinetic and Pharmacogenomic Study of Patients With High-Grade Gliomas Receiving Daily Radiation Therapy and Temozolomide
Brief Title: Pharmacokinetics in Patients With Newly Diagnosed High-Grade Glioma Receiving Temozolomide and Radiation Therapy
Status: Terminated | Type: Observational
Why Stopped: low accrual
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: J0684; P30CA006973 (NIH); CDR0000543866; NA_00004964 (Other: JHM IRB)
Record Dates: First submitted 2007-05-08; First posted 2007-05-10 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Brain and Central Nervous System Tumors; Thrombocytopenia
Keywords: thrombocytopenia; adult anaplastic oligodendroglioma; adult brain stem glioma; adult mixed glioma; adult giant cell glioblastoma; adult gliosarcoma; adult glioblastoma; adult anaplastic astrocytoma; adult anaplastic ependymoma; adult pineal gland astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Thrombocytopenia; Oligodendroglioma; Glioma; Glioblastoma; Gliosarcoma; Astrocytoma; Ependymoma | interventions — Temozolomide; Comparative Genomic Hybridization; Amplified Fragment Length Polymorphism Analysis; Radiotherapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: temozolomide
Genetic: comparative genomic hybridization
Genetic: polymorphism analysis
Other: laboratory biomarker analysis
Other: pharmacological study
Radiation: radiation therapy

SUMMARY:
RATIONALE: Studying samples of blood in the laboratory from patients receiving temozolomide may help doctors learn how temozolomide works in the body. It may also help doctors learn more about how a patient's genes may affect the risk of developing thrombocytopenia.

PURPOSE: This clinical trial is studying the pharmacokinetics in patients with newly diagnosed high-grade glioma receiving temozolomide and radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the pharmacokinetic (PK) profiles of temozolomide (TMZ) in patients who develop severe thrombocytopenia vs PK profiles in patients who do not develop severe thrombocytopenia while receiving standard first-line therapy for management of newly diagnosed high-grade gliomas.
* Determine if patients who develop thrombocytopenia have any single nucleotide polymorphisms in the O6-methylguanine-DNA methyltransferase gene.

OUTLINE: This is a pilot, prospective, multicenter study.

Patients receive oral temozolomide once daily on days 1-42. Patients also undergo cranial radiotherapy 5 days a week for 6 weeks in the absence of disease progression or unacceptable toxicity.

Blood samples are collected periodically for pharmacokinetic and pharmacogenomic analysis, genotype analysis, plasma temozolomide levels, and MGMT repair gene polymorphism analysis.

After completion of study treatment, patients are followed for 1 month.

PROJECTED ACCRUAL: A total of 150 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed high-grade glioma (WHO grade III or IV)
* Must be scheduled to receive standard first-line therapy (cranial radiotherapy and temozolomide)

PATIENT CHARACTERISTICS:

* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 1.7 mg/dL
* Bilirubin ≤ 1.5 mg/dL
* Transaminases ≤ 4 times upper limit of normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except curatively treated carcinoma in situ or basal cell carcinoma of the skin

PRIOR CONCURRENT THERAPY:

* No prior hormonal therapy for brain tumor
* No prior biological agents (including immunotoxins, immunoconjugates, antisense agents, peptide receptor antagonists, interferons, interleukins, tumor-infiltrating lymphocytes, lymphokine-activated killer cells, or gene therapy)
* No prior immunotherapy
* No prior chemotherapy
* No prior radiotherapy, including cranial radiotherapy
* Concurrent glucocorticoid therapy allowed
* No concurrent carbamazepine
* No other concurrent experimental therapy
* No other concurrent cytotoxic therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High grade glioma
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2006-11-11 (Actual); Primary Completion 2008-11-12 (Actual); Study Completion 2009-08-18 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of temozolomide (TMZ) in patients with severe thrombocytopenia after standard first-line therapy as measured by Area Under the Curve (AUC) | Day 1, Day 22, Day 43
  AUC (mg*h/L)in patients who develop severe thrombocytopenia after receiving standard first-line therapy of temozolomide (TMZ) for management of newly diagnosed high-grade gliomas.
Pharmacokinetics (PK) of temozolomide (TMZ) in patients with severe thrombocytopenia after standard first-line therapy as measured by maximum drug concentration (Cmax) | Day 1, Day 22, Day 43
  Cmax in patients who develop severe thrombocytopenia after receiving standard first-line therapy of temozolomide (TMZ) for management of newly diagnosed high-grade gliomas.
Pharmacokinetic (PK) profile of temozolomide (TMZ) in patients without severe thrombocytopenia after standard first-line therapy as measured by AUC | Day 1, Day 22, Day 43
  AUC in patients in patients who do not develop severe thrombocytopenia after receiving standard first-line therapy of TMZ for management of newly diagnosed high-grade gliomas.
Pharmacokinetic (PK) profile of temozolomide (TMZ) in patients without severe thrombocytopenia after standard first-line therapy as measured by Cmax | Day 1, Day 22, Day 43
  Cmax in patients in patients who do not develop severe thrombocytopenia after receiving standard first-line therapy of TMZ for management of newly diagnosed high-grade gliomas.

SECONDARY OUTCOMES:
Presence of single nucleotide polymorphisms in the O6-methylguanine-DNA methyltransferase gene. | Day 1
  Presence of single nucleotide polymorphisms in the O6-methylguanine-DNA methyltransferase gene of patients who develop thrombocytopenia after receiving standard first-line therapy for management of newly diagnosed high-grade gliomas.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A. Grossman, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (2):
- United States (2):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland